CLINICAL TRIAL: NCT04588883
Title: Strengthening Families Living With HIV in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-0241
Record Dates: First submitted 2020-09-15; First posted 2020-10-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: ART; Hiv; Trust; Depression, Anxiety; PTSD; Adherence, Medication
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Patients, adults and adolescents, will be recruited from patient registries at 7 government operated HIV clinics in Meru County, Kenya. Patients will complete validated questionnaires at baseline, 1.5 year and 3 years into a novel adaptation of a community empowerment program. The program utilizes savings- and internal-lending/group-based microfinance process to facilitate exchange of savings amongst patients and adolescent guardians. A byproduct of this process is the development of social capital, which will be used to facilitate education, peer learning, and collective problem solving to improve determinants of well-being and clinical adherence among participants. Expected outcomes include improved viral suppression, ART adherence, clinical attendance, and mental health.
  Interventions: Behavioral: Kuja Pamoja - HIV

INTERVENTIONS:
Behavioral: Kuja Pamoja - HIV — Information has been provided in the treatment arm description.

SUMMARY:
This study seeks to use a group-based microfinance/internal lending model to develop social capital among people with HIV in Kenya. This will create a context to deliver validated curriculum targeting intimate partner violence, positive parenting, agriculture, small business entrepreneurship, group-interpersonal therapy, and other determinants of well-being and ART adherence among people with HIV. The primary outcomes are viral suppression, ART adherence, and common mental disorders.

DETAILED DESCRIPTION:
It is anticipated that involvement in an internal savings and lending program will create social capital among people with HIV and their guardians (in case of adolescents w HIV). This social capital accrual will be leveraged to support and disseminate social skills (i.e. positive parenting, conflict resolution), economic skills (i.e. entrepreneurship, farming), and health skills (i.e. ART adherence, retention in care to produce viral suppression). The overall outcome is improved social, health, and economic well-being.

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion of subjects include:

* testing positive for HIV, confirmed by the Ministry of Health clinics
* being at or older than 13 years of age
* initiating care at a qualified Ministry of Health clinic in the catchment area, or intending to initiate care at such a clinic (see below for definition)
* Any gender, age (13+ years), and comorbid disease states
* Provide informed consent if adult, emancipated minor or mature minor
* Provide assent if minor with guardian, who must provide informed consent

Qualified clinical locations include

* those with accessible and usable public land to convene weekly meetings,
* no current program targeting families with HIV known to the Ministry of Health

Exclusion Criteria:

* Refusal to participate
* Current participation in a similar program
* Residing in a location with a similar program targeting patients with HIV
* Not covered by inclusion criteria.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Viral Suppression | Change from baseline to 3 years
  Viral suppression is measured as an undetectable viral load using standard clinic procedures.
Anti-retroviral therapy Adherence | Change from baseline to 3 years
  Anti-retroviral therapy (ART) adherence will be measured by patient report using the adherence portions of the AIDS Clinical Trial Group (ACTG) Adherence tool and by refill history.
Depression | Change from baseline to 3 years
  Depression will be measured using the Beck's Depression Inventory. Higher scores mean more depressive symptoms present.
Anxiety | Change from baseline to 3 years
  Anxiety will be measured using the Generalized Anxiety Disorder (GAD7) instrument. Higher score means more anxiety symptoms present.
Post-Traumatic Stress Disorder | Change from baseline to 3 years
  Post-traumatic stress disorder (PTSD) will be measured using the PTSD symptom scale. Higher scores mean more PTSD symptoms present.

SECONDARY OUTCOMES:
Group entitativity | Change from baseline to 3 years
  Social cohesion (operationalized as group entitativity) will be measured using the Generalized Entitativity Measure (GEM). Higher score on this visual analogue scale means higher group entitativity.
Intimate partner violence | Change from baseline to 3 years
  Family violence will be measured using the Conflict Tactics Scale (CTS-2). Higher scale scores mean more conflict present; higher violence/coercive subscale scores mean more violence and coercion present.
Food insecurity | Change from baseline to 3 years
  Food security will be measured using the Household Food Insecurity Scale instrument. Higher scale scores mean higher food insecurity.
Social trust | Change from baseline to 3 years
  Social trust will be measured using a single validated item. This is a binary outcome with 1=presence of trust between respondent and other similar aged people with HIV.
Expectations of mutual support | Change from baseline to 3 years.
  Expectation of mutual support will be measured using the a single validated item. Higher score means higher expectation of mutual support between respondent and other similar-aged people with HIV.
Child-guardian conflict | Change from baseline to 3 years.
  Child-guardian conflict will be measured using the Conflict Tactics Scale for children (CTS2-pc). Higher scale score means more conflict present; higher violence subscale scores mean more violent conflicts used.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Goodman, DrPH, Principal Investigator — The University of Texas Medical Branch, Galveston; Stanley Gitari, MPH, Study Director — Sodzo Kenya
Locations (1):
- Meru County Department of Health, Maua, Meru County, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made openly available following acceptance for publication of all main analyses.
Supporting Information: Analytic Code
Time Frame: Data will be available following publication of baseline, 1.5 year and 3 year data panels.
Access Criteria: Interested researchers must send requests to corresponding author, including study questions, statistical plan for analysis and evidence of competence in performing proposed statistical tests.

REFERENCES:
- [Result] Foa, E. B., Riggs, D. S., Dancu, C. V., & Rothbaum, B. O. (1993). Reliability and validity of a brief instrument for assessing post-traumatic stress disorder. Journal of traumatic stress, 6(4), 459-473.
- [Result] Gaertner, L., & Schopler, J. (1998). Perceived ingroup entitativity and intergroup bias: An interconnection of self and others. European Journal of Social Psychology, 28(6), 963-980.
- [Result] Chesney MA, Ickovics JR, Chambers DB, Gifford AL, Neidig J, Zwickl B, Wu AW. Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: the AACTG adherence instruments. Patient Care Committee & Adherence Working Group of the Outcomes Committee of the Adult AIDS Clinical Trials Group (AACTG). AIDS Care. 2000 Jun;12(3):255-66. doi: 10.1080/09540120050042891. PMID 10928201
- [Result] Straus, M. A., Hamby, S. L., Boney-McCoy, S., & Sugarman, D. B. (1996). The revised conflict tactics scales (CTS2) development and preliminary psychometric data. Journal of family issues, 17(3), 283-316.
- [Result] Knack, S., and Keefer, P. (1997) Does social capital have an economic payoff? A cross-country investigation. The Quarterly Journal of Economics, 112(4), 1251-1288.
- [Result] Poortinga W. Social relations or social capital? Individual and community health effects of bonding social capital. Soc Sci Med. 2006 Jul;63(1):255-70. doi: 10.1016/j.socscimed.2005.11.039. Epub 2006 Jan 19. PMID 16427171
- [Result] Straus MA, Hamby SL, Finkelhor D, Moore DW, Runyan D. Identification of child maltreatment with the Parent-Child Conflict Tactics Scales: development and psychometric data for a national sample of American parents. Child Abuse Negl. 1998 Apr;22(4):249-70. doi: 10.1016/s0145-2134(97)00174-9. PMID 9589178